CLINICAL TRIAL: NCT01868503
Title: Phase II Study to Investigate Concurrent Lapatinib and Radiotherapy in Locally Advanced or Locally Recurrent Breast Cancer and the Impact on Breast Cancer Stem Cells
Brief Title: Lapatinib Ditosylate and Radiation Therapy in Treating Patients With Locally Advanced or Locally Recurrent Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Protocol modification
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kathleen Horst, Assistant Professor of Radiation Oncology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRS0027; NCI-2013-01065 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA124435 (NIH)
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lapatinib Plus Radiation Therapy (Experimental): Patients receive lapatinib ditosylate PO QD on day 1 until completion of radiation therapy. Beginning on day 7, patients undergo radiation therapy for 5-7 weeks and will have their blood banked for laboratory biomarker analysis.
  Interventions: Drug: lapatinib ditosylate; Radiation: radiation therapy; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lapatinib ditosylate — Given PO
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well lapatinib ditosylate and radiation therapy work in treating patients with locally advanced or locally recurrent breast cancer. Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x rays to kill tumor cells. Giving lapatinib ditosylate together with radiation therapy may be an effective treatment for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the clinical complete response rate (CR) after concurrent lapatinib (lapatinib ditosylate) and radiotherapy in patients with locally advanced or locally recurrent breast cancer that is refractory to chemotherapy.

SECONDARY OBJECTIVES:

I. To evaluate the feasibility of assessing breast cancer stem cells (BCSCs) using flow cytometry and single cell gene expression profiling (SCGEP).

II. To determine the change in the proportion of BCSCs after combined modality therapy.

III. To evaluate the safety and efficacy of the combination of lapatinib and radiotherapy.

IV. To assess the pathologic complete response rate (pCR) in those undergoing surgical resection.

OUTLINE:

Patients receive lapatinib ditosylate orally (PO) once daily (QD) on day 1 until completion of radiation therapy. Beginning on day 7, patients undergo radiation therapy for 5-7 weeks.

After completion of study treatment, patients are followed up at 2-4 weeks and then at 6-12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed locally advanced breast cancer that is refractory to chemotherapy or other therapeutic agents or with a history of breast cancer with new evidence of a local recurrence (defined as a chest wall or breast recurrence and/or nodal recurrence); the diagnosis will be made based on clinical and pathologic features
* Patients must be >18 years of age.
* Karnofsky Performance Status (KPS) score > 70
* Patts must have normal organ function as defined below:

  * total bilirubin < 1.5 x institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) < 2.5 x institutional upper limit of normal
  * creatinine < 1.5 x institutional upper limit of normal
* Patients must have left-ventricular ejection fraction > 50% at baseline.

Exclusion Criteria:

* Patients who have contraindications to radiotherapy, such as scleroderma, dermatomyositis, or severe cutaneous manifestations of systemic lupus erythematosus (SLE)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lapatinib
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, or psychiatric illness/social situations that would limit compliance with study requirements
* Women who are pregnant or lactating, as well as women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Horst, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University Cancer Institute, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Lapatinib Ditosylate, Radiation Therapy): Patients receive lapatinib ditosylate PO QD on day 1 until completion of radiation therapy. Beginning on day 7, patients undergo radiation therapy for 5-7 weeks.
  lapatinib ditosylate: Given PO
  radiation therapy: Undergo radiation therapy
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Lapatinib Ditosylate, Radiation Therapy)
Started | 7
Completed | 5
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Lapatinib Ditosylate, Radiation Therapy)
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving Complete Clinical Response
Description: Complete clinical response will be defined as the absence of tumor on the chest wall, in the treated breast, or in the nodal regions as assessed by clinical examination +/- radiographic imaging (if clinically indicated).
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib Plus Radiation Therapy
Number analyzed (Participants) | 7
Participants | 2

2. Secondary Outcome: Feasibility of Assessing the Effects of Lapatinib and Radiation Therapy on BCSCs Using Flow Cytometry and SCGEP
Description: Defined as the percentage of biopsy specimens for which the SCGEP assay achieves a non-zero number.
Time Frame: 12 weeks
Population: Data were not collected and the outcome measure was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in the Proportion of BCSCs
Description: Defined as the difference between the percentage of BCSCs before and after treatment. Proportion of biopsy samples that are evaluable for BCSCs will be estimated along with 95% exact confidence intervals. BCSC results will be summarized using medians and interquartile ranges. Changes in BCSCs will be assessed using the Wilcoxon signed rank test.
Time Frame: Baseline to 12 weeks
Population: This outcome was not analyzed due to lack of funding. It may be re-evaluated in the future. Data were not collected and the outcome measure was not analyzed.
Arm/Group | Treatment (Lapatinib Ditosylate, Radiation Therapy)
Number analyzed (Participants) | 0

4. Secondary Outcome: Incidence of Adverse Events Graded According to Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: Adverse events will be tabulated by organ system and severity.
Time Frame: Up to 12 weeks
Population: Participants enrolled in the study.
Measure: Number; unit: incidencts
Arm/Group | Treatment (Lapatinib Ditosylate, Radiation Therapy)
Number analyzed (Participants) | 7
incidencts
  Grade 3 Events | 2
  Grade 4 Events | 1

5. Secondary Outcome: Pathologic Complete Response Rate for Those Patients Undergoing Surgical Resection Defined as no Evidence of Residual Tumor in the Breast and Lymph Nodes
Description: Proportion of patients who achieve a pathological complete response will be estimated with 95% exact confidence intervals.
Time Frame: Up to 12 weeks
Population: Of the patients in the treatment arm, only 1 received surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Lapatinib Ditosylate, Radiation Therapy)
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Lapatinib Ditosylate, Radiation Therapy)
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lapatinib Ditosylate, Radiation Therapy) (N=7)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Fever-Possible sepsis (Infections and infestations) | 1 (1)
Chest Pain (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lapatinib Ditosylate, Radiation Therapy) (N=7)
Alanine aminotransferase increased (Endocrine disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No